CLINICAL TRIAL: NCT07117136
Title: Real World Outcomes of Blinatumomab Consolidation in Patients With B-cell Acute Lymphoblastic Leukemia
Brief Title: Blinatumomab Consolidation in Real World
Status: Recruiting | Type: Observational
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Ehab L Atallah, Assistant Professor, Medical College of Wisconsin
Other Study IDs: PRO00054269
Record Dates: First submitted 2025-08-05; First posted 2025-08-12 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: B-Cell Acute Lymphoblastic Leukaemia
MeSH Terms: conditions — Burkitt Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients who received Blinatumomab Therapy
- Patients who did not receive Blinatumomab Therapy

SUMMARY:
This will be a multi-center registry for patients with B-ALL. Patient data will be collected both retrospectively and prospectively. The data forms and surveys will be built and managed through REDCap, a secure web application managed by the Clinical & Translational Science Institute.

DETAILED DESCRIPTION:
B-cell Acute lymphoblastic leukemia (B-ALL) is a potentially curable malignancy in the pediatric population. In contrast, the outcomes of adults with B-ALL have remained historically poor due to risk of relapse after frontline therapy. Novel agents in the current era have changed the treatment landscape of adults with relapsed/refractory B-ALL with improved tolerability and better outcomes [1]. Currently, blinatumomab (CD3-CD19 bispecific molecule) and inotuzumab (CD22 antibody drug conjugate) are approved for the management of patients with relapsed/refractory B-ALL. With the superior efficacy of these agents, recent clinical trials have focused on incorporating them in the management of newly diagnosed B-ALL.

A phase 3 randomized clinical trial (E1910) has recently demonstrated the superiority of adding blinatumomab during consolidation for patients who have achieved MRD negative CR [2]. Patients between the ages of 30 and 70 with newly diagnosed BCR-ABL1 negative B-ALL were enrolled and initially received 2.5 months of combination induction chemo utilizing a BFM-like regimen adapted from the E2993/UKALLXII clinical trial with extended remission induction, addition of pegasparginase for patients <55 years of age and addition of rituximab for CD20 positive patients. Subsequently, their remission and MRD status were determined centrally by 6-color flow cytometry with MRD negativity defined as <0.01%. All patients were then randomized to receive an additional four cycles of consolidation chemo or two cycles of blin for 28 days each cycle followed by 3 cycles of consolidation chemo, another 4-week cycle of blinatumomab (3rd cycle of blinatumomab) followed by an additional cycle of chemo and then a 4th cycle of blinatumomab. Two hundred and twenty-four MRD negative patients were randomized, 112 pts to each arm. Among the MRD negative patients, superior overall survival was seen in patients who received blinatumomab (median OS: not reached vs. 71.4 months; Hazard ratio 0.42, 95% CI: 0.24 - 0.75; two-sided p=0.003) with a median follow-up of 43 months.

While the results are encouraging and practice changing to consider adding blinatumomab to MRD negative CR patients, the backbone chemotherapy regimen used in E1910 study is not a commonly used regimen in clinical practice. Due to the unmet need, physicians are often considering combining blinatumomab consolidation with several other commonly used chemotherapy regimens. However, the outcome in this setting remains unknown. Our goal in this study is to evaluate the real-world utilization of blinatumomab in the frontline setting for management of B-ALL in the United States.

ELIGIBILITY:
Inclusion Criteria:

* 1) aged 18 years or older 2) diagnosed with B-ALL on or after December 1st 2023 3) Not received blinatumomab in an interventional clinical trial setting 4) Willing and able to give informed consent (or retrospective data for deceased patients

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with B-ALL diagnosed during or after December 2022
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-08-28 (Actual); Primary Completion 2029-05-14 (Estimated); Study Completion 2029-05-14 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with complete remission | 5 years or e.g., 1 year after closure of study
  Complete remission as defined by patients having no lymphoblasts in the marrow or blood

SECONDARY OUTCOMES:
Overall Survival | 5 years
  Percentage of participants overall survival (OS). OS will be calculated from the time of diagnosis of to death from any cause, and patients will be censored if they were alive at the last follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No